CLINICAL TRIAL: NCT04693949
Title: Effect of Nano-structured Alumina Coating on the Bond Strength of Zirconia Resin-bonded Fixed Dental Prostheses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Adhesion of RBFDPs
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Missing Incisors; Zirconia Surface Pretreatment; Children; Adults; Debonding
Keywords: Airborne particle abrasion; Nanostructured alumina coating; Resin-bonded fixed dental prostheses

STUDY DESIGN:
Intervention Model Description: This is a single-centre, prospective, randomized, controlled, double-blind clinical trial.
Who Masked: Participant, Care Provider
Masking Description: Prior to the beginning of the study 50 identification numbers were divided into 2 groups on the basis of a computer generated tables (www.randomization.com). The two groups were then randomly allocated to the zirconia pretreatment method using a random generator. The randomization process was conducted by a staff member not involved in the research protocol. For each identification number, the selected pretreatment is written on a card contained in an opaque sealed envelope. The envelopes are stored by a study supervisor. Each envelope is opened by a dental technician after the RBFDP's zirconia framework is milled and then once again stored by the study supervisor until the conclusion of a study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APA (Active Comparator): Air-borne particle abrasion of zirconia RBFDPs prior to bonding
  Interventions: Other: APA
- NAC (Experimental): Pretreatment of zirconia RBFDP with nanostructured alumina coating after milling of RBFDP's framework
  Interventions: Other: NAC

INTERVENTIONS:
Other: NAC — Pretreatment of zirconia RBFDP with nanostructured alumina coating after milling of RBFDP's framework
  Arms: NAC
Other: APA — Air-borne particle abrasion of zirconia RBFDPs prior to bonding
  Arms: APA

SUMMARY:
The purpose of this study is to evaluate the clinical outcome of resin-bonded fixed dental prostheses (RBFDPs) pretreated with nanostructured alumina coating (NAC).

The study adopts a prospective, randomized, controlled, double-blind design contrasting the use of NAC to air-borne particle abrasion (APA) (control) as a surface pretreatment method of zirconia RBFDPs used for replacing missing central or lateral incisors. The primary outcome evaluated is the retention/survival of the zirconia RBFDPs pretreated with APA and NAC.

DETAILED DESCRIPTION:
Zirconia resin-bonded fixed dental prostheses (RBFDPs) have been regarded as a promising minimally invasive alternative for the replacement of missing central and lateral incisors, offering several advantages to orthodontic space closure or tooth replacement with implant-supported restorations. Debonding of the zirconia RBFDPs represents the main technical complication since clinically established airborne particle abrasion (APA) of an inert zirconia surface does not always provide sufficient resin-bond strength. Further, APA can also impair the mechanical properties of zirconia restoration affecting its long-term success. Nano-structured alumina coating (NAC) presents an alternative non-invasive zirconia surface pretreatment. The aim of this randomized controlled clinical trial is to study the effect of NAC coated bonding surface of zirconia RBFDPs affecting its debonding and clinical survival rate.

The study adopts a prospective, randomized, controlled, double-blind design contrasting the use of NAC to air-borne particle abrasion (APA) as a surface pretreatment method of zirconia RBFDPs. Healthy patients in need of a missing central or lateral incisor replacement are screened and rated to be eligible by two calibrated dentists. RBFDPs are randomly allocated into two groups and inserted by the same operator. The first group, where the bonding surface is pretreated with APA serves a control group. In the second group the restorations are pretreated with NAC. The participants and the operator are blinded to the group assignment in a double-blinded trial design. The primary outcome evaluated is the retention/survival of the RBFDP. Non-parametric tests and Kaplan-Meyer analysis will be used to determine differences between both study groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing central or lateral incisor

Exclusion Criteria:

1. inadequate edentulous space for the pontic
2. signs of bruxism
3. abutment tooth with active periodontal or periapical disease
4. inadequate enamel bonding surface of the abutment tooth
5. inadequate interocclusal space for a retainer wing and a proximal connector
6. pontic guidance
7. physical or psychological disease likely to interfere with normal conduct of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate of zirconia RBFDPs | From baseline through study completion, an average of 1 year
  Survival rate is defined by debonding or restoration loss

SECONDARY OUTCOMES:
Porcelain chipping | From baseline through study completion, an average of 1 year
  Porcelain chipping
Zirconia framework fracture | From baseline through study completion, an average of 1 year
  Zirconia framework fracture
Gingivitis | From baseline through study completion, an average of 1 year
  Visual and tactile inspection of gingiva
Parodontitis | From baseline through study completion, an average of 1 year
  Gingival sulcus depth measurement
Marginal leakage | From baseline through study completion, an average of 1 year
  Discoloration of a restoration margin
Secondary caries | From baseline through study completion, an average of 1 year
  Caries between the tooth and restoration margin

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty - University of Ljubljana Ljubljana, Ljubljana, Slovenia